CLINICAL TRIAL: NCT01823380
Title: Influence of the Vitamin D Blood Levels on the Amyotrophic Lateral Sclerosis Phenotype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8987
Record Dates: First submitted 2013-03-22; First posted 2013-04-04 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis; Vitamin D; Blood Levels
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amyotrophic lateral sclerosis (Other): Blood test
  Interventions: Procedure: Blood test

INTERVENTIONS:
Procedure: Blood test — Blood test

SUMMARY:
The main objective of this study is to investigate the correlation between the rate of motor decline and blood levels of Vitamin D total. Secondary objectives are to investigate the relationship between blood levels of vitamin D and total disease duration of ALS, forced vital capacity, weight loss, age of onset and the start site of ALS.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis is one of the most serious neurodegenerative disease, leading to death in 3 years by progressive paralysis of 4 limbs, speech, swallowing and breathing, and due to a progressive death of central and peripheral neurons. The cause of the disease is unknown, but an immunologically factor is more precisely suspected in ALS. Since 2008, the work of Immunology have shown that vitamin D was a major regulator of immunity. It regulates particularly the function of dendritic cells and regulates the immune response in macrophages. A vitamin D deficiency will induce activation of microglia. In neurology, vitamin D deficiency is associated with a greater impairment in neuronal function. This deficit is associated with a faster alteration of the microvasculature, alteration known to increase neuronal suffering and to enhance the neurodegenerative processes. The investigators postulate that ALS patients have a more severe prognosis if their vitamin D levels at the time of diagnosis is lower. The main objective of this study is to investigate the correlation between the rate of motor decline and blood levels of Vitamin D total. Secondary objectives are to investigate the relationship between blood levels of vitamin D and total disease duration of ALS, forced vital capacity, weight loss, age of onset and the start site of ALS.

ELIGIBILITY:
Inclusion Criteria:

* Subject with possible, probable or definite Amyotrophic Lateral Sclerosis (ALS).
* ALS operating for less than three years at dosage of vitamin D time.
* Subject monitored in the center ALS of Montpellier for 6 months.
* Subject agreeing to give his consent in writing or orally if the patient SLA is unable to write

Exclusion Criteria:

* Subject has received a Vitamine D treatment in the six months preceding the inclusion
* Subject with a clinical condition on the inclusion day that makes it highly probable death in the year (quadriplegic patient, subject ventilated for respiratory failure in ALS, major malnutrition) or with ALSFRS-R score <20.
* Pregnant or breastfeeding women
* Subject not covered by a social security scheme.
* Subject under guardianship
* Adult protected by the law

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2012-09; Primary Completion 2014-02 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Vitamin D blood level | Day 1
  The vitamine D blood level will be assessed the day of the inclusion of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: William Camu, PU PH, Principal Investigator — UH Montpellier
Locations (1):
- UH Montpellier, Montpellier, France